CLINICAL TRIAL: NCT04479800
Title: A Phase 1, Three-Way Crossover Study to Evaluate the Effect of Food on the Pharmacokinetics of ASTX660 in Healthy Volunteers
Brief Title: Effect of Food on the Pharmacokinetics of ASTX660 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: ASTX660-11
Record Dates: First submitted 2020-07-17; First posted 2020-07-21 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — ASTX-660

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment A - Fasting (Experimental): No food prior to dosing
  Interventions: Drug: ASTX660
- Treatment B - Fed (Experimental): High-fat/high-calorie meal prior to dosing
  Interventions: Drug: ASTX660
- Treatment C - Fed (Experimental): Low-fat/low-calorie meal prior to dosing
  Interventions: Drug: ASTX660

INTERVENTIONS:
Drug: ASTX660 — Form: capsule; Route of administration: oral

SUMMARY:
This is a Phase 1, single-dose, open-label, randomized, three-period, three-way crossover study in which healthy adult participants will receive three separate single-dose administrations of ASTX660 capsules under three different conditions.

DETAILED DESCRIPTION:
Participants receiving Treatment A (fasting) will be dosed after having fasted overnight for at least 10 hours. Participants receiving Treatment B (fed; high-fat/high-calorie meal) will fast overnight for at least 10 hours then consume a Food and Drug Administration (FDA) standard high-fat, high-calorie breakfast beginning 30 minutes before dosing. Participants receiving Treatment C (fed; low-fat/low-calorie meal) will fast overnight for at least 10 hours then consume an FDA standard low-fat, low-calorie breakfast beginning 30 minutes before dosing. The duration of the study is expected to be approximately 47 days.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily consents to participate in this study and provides written informed consent before the start of any study-specific procedures.
2. Male or female.
3. Is between 18 and 55 years of age (inclusive).
4. Has a body mass index (BMI) between 18 and 32 kg/m2 (inclusive) and weighs a minimum of 50 kg.
5. Females must be of non-childbearing potential (defined as surgically sterile [i.e. had a bilateral tubal ligation, hysterectomy, or bilateral oophorectomy at least 6 months before the first dose of study medication] or postmenopausal for at least 1 year before the first dose of study medication).
6. Is willing and able to remain in the study unit for the entire duration of the confinement period.
7. Is willing and able to consume the entire FDA standard high-fat and low-fat meal in the timeframe required during the designated study periods.
8. Has vital signs (measured sitting after a minimum 3 minutes rest) at screening within the following ranges: heart rate: 40-100 bpm; systolic blood pressure (BP): 90-145 mmHg; diastolic BP: 50-95 mmHg. Out-of-range vital signs may be repeated once at the Investigator's discretion.

Exclusion Criteria:

1. History or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, oncologic, autoimmune, or psychiatric disease or any other condition that, in the opinion of the Investigator, would jeopardize the safety of the participant or the validity of the study results.
2. A clinically significant abnormal finding on the physical exam, medical history, electrocardiogram (ECG), or clinical laboratory results at screening.
3. Has laboratory values that are not within normal limits for amylase and lipase, phosphorus, alkaline phosphatase (ALP), aspartate transaminase (AST), alanine transaminase (ALT), bilirubin, white blood cell count (WBC) and absolute neutrophil count (ANC), international normalized ratio (INR), C-reactive protein (CRP), or has any other clinically significant abnormal chemistry values in the opinion of the Investigator.
4. Has an ECG parameter (confirmed by repeat evaluation) of PR ≥ 200 ms, or QRS ≥ 110 ms, or QT interval corrected by the method of Fridericia (QTcF) > 450 ms at screening visit.
5. History or presence of allergic or adverse response to ASTX660 or related drugs or ASTX660 excipients.
6. Has been on a significantly abnormal diet (i.e., low-calorie, vegan, or intermittent fasting) during the 4 weeks preceding the first dose of study medication.
7. Has participated in another clinical trial (randomized participants only) within 30 days before the first dose of study medication.
8. Use of any over-the-counter (OTC) medication (including nutritional or dietary supplements, herbal preparations, or vitamins) within 7 days before the first dose of study medication until the end of study visit without evaluation and approval by the Investigator.
9. Use of any prescription medication, except hormonal replacement therapy, from 14 days before the first dose of study medication until the end-of-study visit without evaluation and approval by the Investigator.
10. Has been treated with any known drugs that are moderate or strong inhibitors/inducers of cytochrome P450 (CYP) enzymes (e.g., barbiturates, phenothiazines, cimetidine, carbamazepine) or known P-gp inhibitors, or is taking any concomitant medication within 30 days before the first dose of study medication.
11. Blood or plasma donation within 30 days before the first dose of study medication until the end-of-study visit. It is recommended that blood/plasma donations not be made for at least 30 days after the end-of-study visit.
12. Smoking or use of tobacco- or nicotine-containing products within 60 days before the first dose of study medication until the end-of-study visit.
13. Engagement in strenuous exercise from 48 hours before the first dose of study medication until the end-of-study visit.
14. Consumption of beverages or foods that contain alcohol, grapefruit, poppy seeds, broccoli, Brussels sprouts, pomegranate, star fruit, char-grilled meat, or caffeine/xanthine from 48 hours before the first dose of study medication until the end-of-study visit. Participants will be instructed not to consume any of the above products; however, allowance for an isolated single incidental consumption may be evaluated and approved by the study Investigator based on the potential for interaction with the study drug.
15. Has any prior history of substance abuse or treatment (including alcohol).
16. Is a female with a positive pregnancy test result.
17. Has a positive urine screen for drugs of abuse (amphetamines, barbiturates, benzodiazepines, cocaine, cannabinoids, opiates) or cotinine.
18. Has a positive test for hepatitis B surface antigen, hepatitis C antibody, or human immunodeficiency virus (HIV) at screening or has been previously treated for hepatitis B, hepatitis C, or HIV infection.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2020-08-25 (Actual); Study Completion 2020-08-25 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameter Cmax | Predose to 72 hours postdose, up to Day 4
  Maximum plasma concentration
Pharmacokinetic parameter Tmax | Predose to 72 hours postdose, up to Day 4
  Time to reach maximum plasma concentration
Pharmacokinetic parameter λz | Predose to 72 hours postdose, up to Day 4
  Observed terminal rate constant
Pharmacokinetic parameter t1/2 | Predose to 72 hours postdose, up to Day 4
  Observed terminal half-life
Pharmacokinetic parameter AUC(0-24h) | Predose to 24 hours postdose, up to Day 4
  Area under the concentration-time curve from time-zero to 24 hours postdose
Pharmacokinetic parameter AUClast | Predose to 72 hours postdose, up to Day 4
  Area under the concentration-time curve from time-zero to the time of the last quantifiable concentration
Pharmacokinetic parameter AUCinf | Predose to 72 hours postdose, up to Day 4
  Area under the concentration-time curve from time-zero extrapolated to infinity
Pharmacokinetic parameter AUCExtrap (%) | Predose to 72 hours postdose, up to Day 4
  Percentage of AUCinf based on extrapolation
Pharmacokinetic parameter Clast | Predose to 72 hours postdose, up to Day 4
  Last quantifiable concentration determined directly from individual concentration-time data
Pharmacokinetic parameter Tlast | Predose to 72 hours postdose, up to Day 4
  Time of the last quantifiable concentration

CONTACTS AND LOCATIONS:
Locations (1):
- Worldwide Clinical Trials, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No